CLINICAL TRIAL: NCT06046534
Title: ERYTHRO Retrospective Medical Chart Review Study to Describe the Experience of SLE Patients Treated With Anifrolumab in the Early Access Programs.
Brief Title: Retrospective Medical Chart Review Study to Describe the Experience of SLE Patients Treated With Anifrolumab in the Early Access Programs.
Acronym: ERYTHRO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: CernerEnviza / Oracle (Unknown)
Responsible Party: Sponsor
Other Study IDs: D3461R00058
Record Dates: First submitted 2023-06-27; First posted 2023-09-21 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: chronic autoimmune disease; immunosuppressants; corticosteroids; human monoclonal antibody (IgG1ƙ mAb); Real World
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: SLE patients who participated in the anifrolumab EAPs (AMANA or ATUc).
  Interventions: Other: None (Observational study)

INTERVENTIONS:
Other: None (Observational study) — Not applicable since this is observational study.

SUMMARY:
The ERYTHRO study is a retrospective medical chart review study of patients in the AMANA and ATUc Early Access Programs (EAPs) across a number of countries, to assess anifrolumab usage and patient experience in treating SLE in a real-world setting. Since patient safety data are already collected and reported according to regulatory requirements through EAPs, this study will not collect safety data.

DETAILED DESCRIPTION:
This is a multi-country, multi-site retrospective chart review study that will use data extracted from the medical charts of SLE patients who participated in the anifrolumab EAPs AMANA or ATUc in France, Germany, Greece, Israel, Italy, Portugal, Spain, and the UK. Patient level data will be captured longitudinally for each patient over a 12- to 18-month period. The study period will include retrospective data collection covering a minimum 6- month baseline period prior to the index date and retrospective data collection covering a minimum 6-month FU period from the first Anifrolumab infusion. The index date is defined as the date of first anifrolumab infusion during the indexing period. The indexing period is between the earliest date of patient enrolment into the EAP and the date of last new patient enrolment into EAP. The EAPs have closed by end of February 2023 in all countries included in the ERYTHRO study. One data extraction will be performed per patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of enrolment into AMANA or France ATUc program, and
* Have at least 6 months of data from medical charts available prior to the initiation of anifrolumab through the EAP, and
* Have been initiated on anifrolumab at least 6 months before enrolment into ERYTHRO study, and
* Informed consent obtained (where required as per country regulations) to participate in ERYTHRO

Exclusion Criteria:

* Participated in anifrolumab clinical trials, NCT02794285 (D3461C00009) and / or NCT01753193 (D3461C00003), prior to enrolment into AMANA or France ATUc program, or
* Participated in any SLE clinical trial during the baseline period and / or the FU period of ERYTHRO, or
* Patients who were pregnant during the baseline period and / or the FU period of ERYTHRO

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is defined as adult SLE patients enrolled in AMANA EAP or the anifrolumab France ATUc and meeting the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Disease activity assessed by Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) or any of its components at 6 months from the date of first anifrolumab infusion | 6-month longitudinal data capture
  The SLEDAI-2K stands for Systemic Lupus Erythematosus Disease Activity Index -2000. It measures disease activity in the 28 days prior to and at the time point of the assessment. It is a global index and includes 24 clinical symptoms and laboratory variables that are weighted by the type of manifestation, but not by severity or dynamic of the individual item. The SLEDAI-2K includes scoring for antibodies (anti-dsDNA positive or negative) and low complement, as well as some renal and hematologic parameters. The total score ranges between 0 and 105, with higher scores representing increased disease activity. In practice it is expected that SLEDAI scores will be skewed towards 0, with scores higher than 20 being rare.
Disease activity assessed by the Physician Global Assessment (PGA) at 6 months from the date of first anifrolumab infusion | 6-month longitudinal data capture
  The PGA is a single-item visual analogue scale that describes the physician assessment of a patient's disease and its impact on daily functioning at the time of assessment. The scale ranges from 0 (asymptomatic disease and no limitation of normal activities) to 3 (severe disease and limitation of normal activities).
  0 - none
  1. - mild
  2. - moderate
  3. - severe

SECONDARY OUTCOMES:
1. Proportion of patients achieving SLE remission at 6 months from the date of first anifrolumab infusion | 6-month longitudinal data capture
  Remission: defined as clinical SLEDAI = 0, and PGA < 0.5. The patients may be on antimalarials, low-dose glucocorticoids (prednisolone ≤ 5 mg/day), and/or stable immunosuppressives, including biologics
2. Proportion of patients achieving all four criteria for low disease activity (LLDAS) at 6 months from first anifrolumab infusion | 6-month longitudinal data capture
  LLDAS assessment requires all of the following criteria to be met:
  1. SLEDAI-2K score ≤ 4, with no activity in major organ systems (renal, central nervous system, cardiopulmonary, vasculitis, or fever),
  2. No new SLEDAI-2K assessed disease activity compared with the previous visit,
  3. PGA score ≤ 1,
  4. Prednisone or equivalent dosage ≤ 7.5 mg/day, and
  5. No non-standard immunosuppressant dosing, with antimalarials allowed.
3. The frequency overall and by intensity (mild / moderate and severe) of flares as assessed by the Revised Safety of Estrogens in Lupus National Assessment - SLE Disease Activity Index Flare Index (rSFI) at baseline and during follow up. | 6-month longitudinal data capture
  Worsening of symptoms, referred to as flares, will be defined based on the the Revised Safety of Estrogens in Lupus National Assessment-Systemic Lupus Erythematosus Disease Activity Index Flare Index (rSFI). Flares will be categorized into mild/moderate and severe flares as per the rSFI definitions.
4. The extent of skin manifestations over time as described by Cutaneous LE Disease Area and Severity Index (CLASI) during baseline and at 6 months after the data of first anifrolumab infusion | 6-month longitudinal data capture
  The Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) consists of 2 scores; the first summarizes the activity of the disease and the second is a measure of the damage done by the disease. Activity is scored on the basis of erythema, scale/hypertrophy of skin and mucous membranes, acute hair loss, and nonscarring alopecia. Damage is scored in terms of dyspigmentation and scarring, including scarring alopecia.
  Study participants are asked whether dyspigmentation due to cutaneous lupus erythematosus lesions usually remains visible for more than 12 months, which is taken to be permanent. If the dyspigmentation lasts longer than 12 months after the active lesion has resolved, then the score is doubled. The scores are calculated by simple addition and range from 0-70 for activity and 0-56 for damage, with higher scores indicating worse disease activity/damage.
5. SLE treatments used before, during and after Anifrolumab, especially oral corticosteroids (OCS) | 12- to 18-month longitudinal data capture
  1. Pre- Anifrolumab treatment/ OCS usage before anifrolumab initiation
  2. Treatment concomitant with Anifrolumab / OCS usage concomitant with Anifrolumab
  3. Post-Anifrolumab treatment/ OCS usage after anifrolumab end/discontinuation.
6. Usage of anifrolumab, including adherence | 12- to 18-month longitudinal data capture
  Adherence is the actual number of infusions received out of the expected number of infusions during a specified duration
7. Usage of anifrolumab, including persistence | 12- to 18-month longitudinal data capture
  Persistence is the time on treatment as per indicated treatment interval
8. Baseline patient characteristics | 12- to 18-month longitudinal data capture
  1. Demographics (age, gender, ethnicity)
  2. Patients medical history
     * Family history of autoimmune diseases
     * Baseline comorbid conditions
     * SLE treatment history
  3. Lifestyle (smoking history, alcohol consumption history)
9. Describe baseline comorbidities described by Charlson Comorbidity Index (CCI) or any of its components | 12- to 18-month longitudinal data capture
  Charlson Comorbidity Index (CCI) predicts the mortality for a patient who may have a range of concurrent conditions, includes 17 chronic diseases in estimating the CCI. The CCI predicts 10- year mortality risk from chronic comorbidities.
10. SLE related tests performed during baseline and FU, respectively | 12- to 18-month longitudinal data capture
  Whole blood tests
11. SLE related tests performed during baseline and FU, respectively | 12- to 18-month longitudinal data capture
  Biochemical
12. SLE related tests performed during baseline and FU, respectively | 12- to 18-month longitudinal data capture
  Serological
13. SLE related tests performed during baseline and FU, respectively | 12- to 18-month longitudinal data capture
  Urine test

CONTACTS AND LOCATIONS:
Locations (15):
- France (6):
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Paris
  - Research Site, Toulouse
- Research Site, Athens, Greece
- Israel (2):
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Research Site, Pisa -PI-, Italy
- Research Site, Porto, Portugal
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Coslada, Madrid
  - Research Site, Valladolid
- Research Site, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3461R00058&attachmentIdentifier=6d51a344-2089-4475-a738-7c8eb3b1edc9&fileName=ERYTHRO_AZ_CSR_Synopsis.pdf&versionIdentifier=